CLINICAL TRIAL: NCT00675818
Title: The Optimal Mode of Renal Replacement Therapy in Acute Kidney Injury (OMAKI) Study: A Pilot Randomized Controlled Trial of Convective Versus Diffusive Clearance
Brief Title: The Optimal Mode of Renal Replacement Therapy in Acute Kidney Injury (OMAKI) Study
Acronym: OMAKI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Ron Wald, Staff Physician/Scientist, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07097
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; renal replacement therapy; critical care unit; hemodialysis; hemofiltration
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CVVH: Patients in this arm will receive CVVH at a replacement fluid rate of 35 mL/kg/h.
  Interventions: Device: Continuous venvenous hemofiltration (CVVH)
- 2 (Active Comparator): CVVHD: Patients in this arm will receive CVVHD at a dialysate flow rate of 35 mL/kg/h.
  Interventions: Device: Continuous venovenous hemodialysis (CVVHD)

INTERVENTIONS:
Device: Continuous venvenous hemofiltration (CVVH) — Continuous venovenous hemofiltration with a replacement fluid rate of 35 mL/kg/hr.
  Arms: 1
Device: Continuous venovenous hemodialysis (CVVHD) — Continuous venovenous hemodialysis at a dialysate flow rate of 35 mL/kg/hr.
  Arms: 2

SUMMARY:
Acute kidney injury (AKI) in the intensive care unit is common, devastating and costly. However, minimal evidence exists to guide the prescription of optimal renal replacement therapy (RRT). An important area of uncertainty surrounds the relative effects of convective versus diffusive modes of clearance. Although both clearance modes provide similar degrees of small molecule clearance, convective modes permit the enhanced clearance of larger-sized molecules which may mediate kidney and systemic toxicity in the setting of AKI.

Continuous renal replacement therapies (CRRTs) are frequently applied in critically ill patients with AKI. Convective clearance, as applied through continuous venovenous hemofiltration (CVVH) and diffusive clearance, as applied through continuous venovenous hemodialysis (CVVHD), may be readily compared in the context of patients receiving CRRT.

The purpose of this study is to examine the feasibility of conducting a larger study that will determine whether convective clearance (hemofiltration) confers improved outcomes as compared to diffusive clearance (hemodialysis) in patients with AKI.

DETAILED DESCRIPTION:
The optimal mode of clearance in critically ill patients with acute kidney injury (AKI) who require renal replacement therapy (RRT) is unclear. Although both convection (as provided by hemofiltration) and diffusion (as provided by hemodialysis) provide equivalent removal of small-sized molecules, hemofiltration offers the potential for removal of large molecules many of which may be toxic. Hemofiltration and hemodialysis have never been compared in a rigorous randomized trial to date.

Continuous renal replacement therapies (CRRT) are widely used in the management of critically ill patients with AKI and current CRRT technology provides a practical platform on which to compare convective and diffusive clearance. We hypothesize that continuous venovenous hemofiltration (CVVH)- at identical doses of small molecule clearance that are provided by the comparison treatment of continuous venovenous hemodialysis (CVVHD)- leads to improved patient outcomes.

This study is an unblinded pilot RCT designed to test the feasibility of conducting a subsequent large scale study that will assess whether CVVH leads to improved patient outcomes (ie, survival, renal recovery) as compared to CVVHD. Although we will be collecting the full array of patient-relevant data for up to 60 days following randomization, the main purpose of this pilot study is to demonstrate the feasibility of recruiting, treating and following patients for a study designed to test this hypothesis.

Patient Population

The recruitment target for this study is 75 patients.

The inclusion and exclusion criteria are designed to enroll patients with AKI on the basis of presumed acute tubular necrosis who would ordinarily be candidates for continuous renal replacement therapies (CRRT) in Canada. The overall philosophy is to enroll and begin applying the study therapy as close as possible to the clinical need to start renal replacement therapy. Similarly, we would like to avoid enrolling patients whose risk of death is so high that the study therapy is unlikely to impact on the clinical outcome.

Treatments

We will employ equivalent doses of hemofiltration (35 mL/kg/hr of replacement fluid) and hemodialysis (35 mL/kg/hr of dialysate).

Therapies will be administered using Primsaflex machines (Gambro Inc.) using regional citrate anticoagulation, heparin anticoagulation or no anticoagulation. Hospital-specific protocols for anticoagulation will be used. We have obtained Health Canada permission to utilize Prismocal, Normocarb, Hemosol BO and Prismasol 4 as infusates in patients receiving CVVH.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (over 16 years of age) admitted to a participating ICU
2. Serum creatinine increase of ≥ 50% from baseline
3. Hemodynamic instability as defined by the cardiovascular component of the SOFA score of ≥ 1
4. Attending physician deems the patient a candidate for RRT for at least one of the following reasons:

   1. Presence of oliguria, defined as a urine output of < 100 mL in the preceding 4 hours
   2. metabolic acidosis (HCO3- < 15 mmol/L and pH < 7.25)
   3. refractory hyperkalemia (K > 6.0 mmol/L)
   4. azotemia (BUN > 50 mmol/L)
   5. suspected uremic organ involvement (pericarditis, encephalopathy, neuropathy or myopathy)

Exclusion Criteria:

1. renal replacement therapy within the previous 2 months
2. presence of renal obstruction
3. receipt of a kidney transplant in the previous year
4. diagnosis of rapidly progressive glomerulonephritis, vasculitis, or acute interstitial nephritis
5. indication for intermittent hemodialysis, specifically severe hyperkalemia, dialyzable drug or toxin
6. terminal illness with associated life expectancy less than 2 months
7. patients who are moribund
8. prior enrollment in this study
9. enrollment in a competing ICU interventional study
10. no CRRT machine available
11. acute renal replacement ongoing for > 36 hours

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
We will study the feasibility of recruiting ther target population, administering the study therapies according to pre-defined protocols and following patients for clinical endpoints. | 60 days

SECONDARY OUTCOMES:
Change in Sequential Organ Failure Assessment (SOFA) score. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wald, MDCM, Principal Investigator — St. Michael's Hospital and University of Toronto
Locations (5):
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Wald R, Friedrich JO, Bagshaw SM, Burns KE, Garg AX, Hladunewich MA, House AA, Lapinsky S, Klein D, Pannu NI, Pope K, Richardson RM, Thorpe K, Adhikari NK. Optimal Mode of clearance in critically ill patients with Acute Kidney Injury (OMAKI)--a pilot randomized controlled trial of hemofiltration versus hemodialysis: a Canadian Critical Care Trials Group project. Crit Care. 2012 Oct 24;16(5):R205. doi: 10.1186/cc11835. PMID 23095370